CLINICAL TRIAL: NCT02116855
Title: Individualized Tertiary Low Dose Prophylaxis for Severe Hemophilia A Children With Arthropathy in China
Brief Title: Individualized Prophylaxis for Severe Hemophilia A Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Runhui WU, Deputy Director of Hematology-Oncology Center, Beijing Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BCH-20140415
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- tertiary prophylaxis prophy on Hemophilia A patiets (Experimental): A multi centre 2 year long term tertiary prophylaxis study designed with a three step escalating dose protocol adjusted by individual joint bleeding patterns/frequencies to study the effect and cost saving of 3 low dose /cost prophylaxis regimens in boys with severe hemophilia A and arthropathy in China. Each patient will start treatment with a low dose regimen in step I and be assessed every 3 months according to the escalating criteria.
  Interventions: Other: according to the efficacy of AJBRs

INTERVENTIONS:
Other: according to the efficacy of AJBRs

SUMMARY:
A multi centre two year long term escalating dose tertiary prophylaxis study on the efficacy and cost saving of individualized low dose prophylaxis regimens for boys with severe hemophilia A in China staring with a low dose regimen in step I, an escalated low dose regimen in step II and a tailored dose regimen based on individual PK profiles in step III. The dose escalation criteria are adjusted according to patterns and frequencies of joint bleeding and assessed in each subject every 3 months. Efficacy of the 3 different dose regimens are measured by the Annualized Joint Bleeding rate (AJBR) as a primary end point and the Hemophilia Joint Health Score (HJHS ) and QoL scores (CHO-KLAT and PedsQoL) , image studies of target joints by Ultrasound, X-ray and MRI examinations, consumption of factor VIII and inhibitor rates as secondary end points.

ELIGIBILITY:
Inclusion Criteria:

1. Severe hemophilia A with FVIII <1 %
2. Age from 6 to 10 years
3. Patients with more than 50 exposure day (ED)
4. Patients with one or more target joints (a target joint is defined as a joint with 3 or more bleeds in a consecutive 3 months) or disease joints (defined as presence of visible joint swelling and /or limitation of movements and/or joint deformities in the absent of an acute joint bleed )
5. on-demand treatment more than 12months before the study

Exclusion Criteria:

1. A history of FVIII inhibitor (titer greater than 0.6 BU) and detectable FVIII inhibitor at screening (titer greater than 0.6 BU)
2. Chronic renal failure (serum creatinine greater than 2.0 mg /dL)
3. Chronic Liver disease (ALT greater than 200 U/L))
4. Patients with clinically documented immunodeficiencies
5. Patients anticipated to require Major surgery
6. Patients with competing high risks such as symptomatic HIV infection, Juvenile rheumatoid arthritis, metabolic bone diseases, or other diseases known to mimic or cause joint diseases
7. Patients live too far from the comprehensive care centre at BCH and had demonstrated previous non compliance to therapies or clinical studies

Ages: 6 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
AJBRs (annualized Joint bleeding rates) | three months

CONTACTS AND LOCATIONS:
Overall Officials: hui R Wu, MD, Study Chair — Beijing Children's Hospital